CLINICAL TRIAL: NCT03244397
Title: Effectiveness of Physical Therapy on Pelvic Organ Prolapse Stages I & II
Brief Title: Physical Therapy on Pelvic Organ Prolapse
Acronym: PT-POP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Maria Torres Lacomba, Professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21/2012
Record Dates: First submitted 2017-08-03; First posted 2017-08-09 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Two groups: Experimental group and Control group
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PT group (Experimental): The participants assigned to this group will receive 16 sessions of physical therapy. Each session will last 45/50 minutes, 2 sessions a week for 8 weeks.
  A directly pelvic floor muscle(PFM) training protocol will be applied. Throw vaginal palpation and in lithotomy position, participants will perform PFM exercises per the treatment proposed by the PERFECT scheme. Biofeedback exercises will be also performed in lithotomy position. Hypopressive exercises which are also home daily from the eighth session. Plus educational strategy.
  Interventions: Other: Physical therapy + educational strategy
- Control group (Active Comparator): Only educational strategy 1 session per week for 6 weeks (every session will last 40/45 minutes). The educational strategy will consist of instruction of printed materials and dimensional anatomical models about the anatomy of the pelvic floor and the physiology of the pelvic organs. It will be recommended to avoid risk factors, such as gaining weight, weight lifting, high impact sports, constipation, smoking, or drinking too much caffeine. They will be also instructed in toilet habits, and will be taught to use the knack maneuver before and during increases of intra-abdominal pressure.
  Interventions: Behavioral: Educational strategy

INTERVENTIONS:
Other: Physical therapy + educational strategy — See arm/group descriptions
  Arms: PT group
Behavioral: Educational strategy — See arm/group descriptions
  Arms: Control group

SUMMARY:
OBJECTIVE: To find out the effectiveness of physical therapy for stages I and II pelvic organ prolapse. DESIGN: Randomized, controlled and single blinded clinical trial. Patients will be randomly assigned to one of these groups: Experimental group: physical therapy + training in lifestyle advice; Control group: just training in means of lifestyle advice. In both groups several physical therapy assessments will be undertaken: 1st before intervention; 2nd immediately after completing intervention; 3rd, 4th, 5th and 6th after 3, 6, 12 and 24 months. SUBJECTS: Women with previously untreated prolapse of stage I or II (confirmed by their gynaecologist using the POP-Q) in Príncipe de Asturias Hospital, provided that there is no contraindication for physical therapy, and after reading, understanding and freely signing an informed consent form. SAMPLE SIZE: A total of 120 subjects will be included in the study (60 subjects in each group). DATA ANALYSIS: A descriptive analysis will be done of all the variables, as well as bivariate analysis in order to find all the possible relationships between the variables. A confidence level of 95% (p<0.05) will be established for all the cases. Effectiveness will be evaluated by comparing between the two groups of the change in outcome variables between visits.

ELIGIBILITY:
Inclusion Criteria:

* Women with POP of any stage I or II according to POP-Q system.

Exclusion Criteria:

* Women diagnosed with POP stage III or IV according to POP-Q system
* Women with a history of conservative POP treatment or surgery
* Women with concomitant disease that may affect treatment (neurological, gynecological or urological) or urinary tract infection or recurrent hematuria
* Women who are pregnant or have had a vaginal birthing the last six months
* Women with cognitive limitations in understanding the information, answer questionnaires, consent and / or participate in the study

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Change of Life impact of Pelvic Floor Dysfunction (PFD) will be assessed by the PFIQ-7 Spanish version. | 6 assessments to evaluate the change from baseline: at baseline, after the intervention period, 3 months, 6 months, 12 months and 24 months after the intervention.
  The PFIQ-7 consists of 3 scales of 7 questions each taken from the Urinary Impact Questionnaire, the Pelvic Organ Prolapse Impact Questionnaire, and the Colorectal-Anal Impact Questionnaire. The 3 scales are scored from 0 (least impact) to 100 (greatest impact) and an overall summary score (0 to 300).
Change of Symptoms and Quality of life (QoL) will be assessed by P-QOL & PFDI-20 Spanish versions | 6 assessments to evaluate the change from baseline: at baseline, after the intervention period, 3 months, 6 months, 12 months and 24 months after the intervention.
  P-QOL assess the symptom severity and its impact on the quality of life in women with POP; and the PFDI-20 that is both a symptom inventory and a measure of the degree of bother and distress (QoL) caused by pelvic floor symptoms. The PFDI-20 includes 20 questions and 3 scales. Each of the 3 scales is scored from 0 (least distress) to 100 (greatest distress). The sum of the scores of these 3 scales serves as the overall summary score of the PFDI-20 and ranges from 0 - 300 and the higher the score, the worse QoL. The 3 scales include questions taken from the following widely used outcome measures: Urinary Distress Inventory - 6 questions, Pelvic Organ Prolapse Distress Inventory - 6 questions, and Colorectal-Anal Distress Inventory - 8 questions collecting data about UI, POP and colorectal and anal symptoms.
Change of Pelvic Floor Muscle (PFM) strength will be measured by manometry | 6 assessments to evaluate the change from baseline: at baseline, after the intervention period, 3 months, 6 months, 12 months and 24 months after the intervention.
  Three maximum PFM contractions will be requested and will be used the mean value. For the manometry (cm2O2), an air-filled probe will be used ("Peritron", Melbourne, Australia)
Change of pelvis floor muscles (PFM) condition by vaginal palpation using Oxford Test | 6 assessments to evaluate the change from baseline: at baseline, after the intervention period, 3 months, 6 months, 12 months and 24 months after the intervention.
  Oxford test range from 0 to 5, according to the muscles strength
Change of Pelvic Floor Muscle (PFM) strength will be measured by dynamometry | 6 assessments to evaluate the change from baseline: at baseline, after the intervention period, 3 months, 6 months, 12 months and 24 months after the intervention.
  Three maximum PFM contractions will be requested and will be used the mean value. For the dynamometry (gr) a two-arms speculum ("Pelvimeter Phenix", Montpellier, France) in mid-sagittal plane, and in close position will be utilized.
Change of pelvis floor muscles (PFM) condition by vaginal palpation Levator Any Test (LAT) | 6 assessments to evaluate the change from baseline: at baseline, after the intervention period, 3 months, 6 months, 12 months and 24 months after the intervention.
  LAT range from 0 to 5, according to the muscles strength and endurance

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Physiotherapy in women´s health research group. University of Alcalà, Alcalà de Henares, Madrid
  - University of Alcalá. FPSM research group. HUPA, Alcalá de Henares, Madrid

IPD SHARING:
Plan to Share IPD: No